CLINICAL TRIAL: NCT00735319
Title: Transcutaneous Bilirubinometers in the Community and the Reduction of Morbidity Associated to Jaundice: A Clustered Randomized Controlled Trial.
Brief Title: Transcutaneous Bilirubinometers in the Community
Acronym: TcB RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other); Capital Health, Canada (Other)
Responsible Party: Dr. Thierry Lacaze, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 7034
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Jaundice, Neonatal
Keywords: Neonatal Jaundice; Physiological Neonatal Jaundice; Neonatal Hyperbilirubinemia; Transcutaneous Bilirubinometer
MeSH Terms: conditions — Jaundice, Neonatal; Hyperbilirubinemia, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (No Intervention): In the 7 control Capital Health community health centers, babies will be followed up according to the current policy. Bilirubin determinations will be performed at the discretion of the visiting nurse if the infant is inappropriately jaundiced or at the request of the physician if risk factors are present. Transcutaneous Bilirubinometers will not be available in each of these 7 centers for all the duration of the study.
- B (Experimental): For all eligible babies living in the 7 intervention community health centers, a Transcutaneous Bilirubinometer will be routinely used by all community nurses in conjunction with an algorithm that will guide the nursing management of the neonates based on the values obtained.Depending on the level of bilirubin obtained and whether risk factors (gestational age < 38 weeks, blood group incompatibility with DAT positive) are present or not, a different management plan will apply. The algorithm is based on curves established by Bhutani et al to predict the risk of significant hyperbilirubinemia based on predischarge bilirubin measurements.
  Interventions: Device: Transcutaneous Bilirubinometer

INTERVENTIONS:
Device: Transcutaneous Bilirubinometer — For all eligible babies living in the 7 intervention community health centers, a Transcutaneous Bilirubinometer will be routinely used by all community nurses in conjunction with an algorithm that will guide the nursing management of the neonates based on the values obtained
  Other Names: Minolta/Drager Air Shields JM-103 Jaundice Meter
  Arms: B

SUMMARY:
Jaundice is the most frequent reason for readmission for healthy newborns after discharge from the nursery. In the Capital Health area, around 2.5% (315 babies in 2005) of all healthy newborns were admitted to the hospital for jaundice. Although jaundice is very common, it is not always a benign condition. If left untreated, it can have devastating consequences including cerebral palsy and hearing loss. It is therefore critical to be able to identify the newborns at risk for severe jaundice. So far, heel puncture of blood collection has been the traditional method to monitor jaundice in newborns. This causes pain to infants, generates anxiety in parents, and consumes significant health care resources. The aim of this study is to evaluate the efficacy of a new and noninvasive screening tool, the transcutaneous bilirubinometer, in detecting babies in our communities who require hospital readmission. This study will demonstrate whether incorporating transcutaneous bilirubinometer in the home care program delivered by nurses of Healthy Beginning allows the early detection of babies at risk of developing severe jaundice at a lower cost and with less discomfort.

ELIGIBILITY:
Inclusion Criteria:

* All near term (35 and 36 weeks gestational age) and term (37 to 41 weeks) babies living in Alberta Capital Health (CH) region
* Born at any Capital Health or Caritas delivery facility(Royal Alexandra Hospital, Grey Nuns Community Hospital, Misericordia Community Hospital, Sturgeon Community Hospital, Fort Saskatchewan Health Centre, and WestView Health Centre)
* Discharged home from the nursery within 96 hours of life

Exclusion Criteria:

* Babies who do not live in CH region
* Babies born at less than 35 weeks gestational age
* Babies initially admitted to a Special Care Nursery (SCN) or a Neonatal Intensive Care unit (NICU) for more than 72 hours
* Babies born to opting-out mothers will also be excluded

Ages: 24 Hours to 2 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10000 (Estimated)
Dates: Start 2008-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Percentage of neonates with at least one serum bilirubin measurement over the 95th percentile, i.e. 350 micromoles/L after 48 hours of age. | From discharge home to 15 days of age

SECONDARY OUTCOMES:
Number of serum bilirubin assessments, number of readmissions, length of admissions, highest level of bilirubin attained, and severity of treatment required | From discharge home to 15 days of age

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Lacaze, MD PhD FRCPC, Principal Investigator — University of Alberta; Philip Etches, MD, Principal Investigator — University of Alberta
Locations (6):
- Canada (6):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Sturgeon Community Hospital, Edmonton, Alberta
  - Fort Saskatchewan Health Centre, Ft Saskatchewan, Alberta
  - WestView Health Centre, Stony Plain, Alberta